CLINICAL TRIAL: NCT02583893
Title: A Biomarker Validation Study to Establish Whether Serial Flow Cytometric Measurements Predict Clinical Response to Sirolimus and MEC (Mitoxantrone Etoposide Cytarabine) Treatment in Patients With High-Risk Acute Myelogenous Leukemia
Brief Title: Biomarkers in Predicting Treatment Response to Sirolimus and Chemotherapy in Patients With High-Risk Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15D.377; 2013-087 (Other: PRC); NCI-2015-01507 (Other: NCI Trial ID)
Record Dates: First submitted 2015-10-08; First posted 2015-10-22 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sirolimus; Mitoxantrone; Etoposide; etoposide phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus, MEC chemotherapy (Experimental): Patients undergo collection of bone marrow samples prior to sirolimus dosing on day 4 and within 1 week and no later than day 45 of hematologic recovery. Patients receive sirolimus PO on days 2-9 (loading dose on day 1 only), and standard MEC chemotherapy comprising mitoxantrone hydrochloride IV over 15 minutes, etoposide IV over 1 hour, and cytarabine IV over 1 hour every 24 hours on day 4-8.
  Interventions: Drug: Sirolimus; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Sirolimus — Given PO
  Other Names: Rapamycin
Drug: Mitoxantrone — Given IV
  Other Names: Mitoxantrone hydrochloride; Novantrone
Drug: Etoposide — Given IV
  Other Names: Etoposide phosphate; VP-16; Etopophos
Drug: Cytarabine — Given IV
  Other Names: Cytosine arabinoside; Cytosar-U; Depocyt; ara-C

SUMMARY:
This pilot phase II trial studies whether biomarkers (biological molecules) in bone marrow samples can predict treatment response to sirolimus and chemotherapy (mitoxantrone hydrochloride, etoposide, and cytarabine [MEC]) in patients with acute myeloid leukemia (AML) that is likely to come back or spread (high-risk). Sirolimus inhibits or blocks the pathway that causes cancer cells to grow. Adding sirolimus to standard chemotherapy may help improve patient response. Studying samples of bone marrow from patients treated with sirolimus in the laboratory may help doctors learn whether sirolimus reverses or turns off that pathway and whether changes in biomarker levels can predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the association between biochemical response and clinical response.

SECONDARY OBJECTIVES:

I. To estimate complete response rate of sirolimus MEC in patients with high risk AML.

II. To estimate progression free survival in this patient population. III. To collect further information on the safety, tolerability, and efficacy of sirolimus in combination with MEC in patients with relapsed or refractory myeloid malignancies.

OUTLINE:

Patients undergo collection of bone marrow samples prior to sirolimus dosing on day 4 and within 1 week and no later than day 45 of hematologic recovery. Patients receive sirolimus orally (PO) on days 2-9 (loading dose on day 1 only), and standard MEC chemotherapy comprising mitoxantrone hydrochloride intravenously (IV) over 15 minutes, etoposide IV over 1 hour, and cytarabine IV over 1 hour every 24 hours on day 4-8.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic evidence of high risk acute myeloid leukemia defined as one of the following:

   1. Primary refractory non-M3 AML

      * Residual leukemia after a minimum of 2 prior courses of chemotherapy (Same or different)
      * Evidence of leukemia recurrence after a nadir bone marrow biopsy demonstrates no evidence of residual leukemia.
      * Evidence of leukemia after induction therapy which, in the opinion of the investigator, would be appropriate for reinduction with sirolimus/MEC therapy.
   2. Relapsed non-M3 AML
   3. Previously untreated non-M3 AML age >60 with no evidence of favorable karyotype defined by presence of t(8;21)(q22;q22) [AML1-ETO], inv16(p13;q22), or t(16;16)(p13;q22) [CBFβ;MYH11] by cytogenetics, FISH, or RT-PCR
   4. Previously untreated secondary AML (from antecedent hematologic malignancy or following therapy with radiation or chemotherapy for another disease) with no evidence of favorable karyotype defined by presence of t(8;21)(q22;q22) [AML1-ETO], inv16(p13;q22), or t(16;16)(p13;q22) [CBFβ;MYH11] by cytogenetics, FISH, or RT-PCR
2. Subjects must be ≥ 18 years of age.
3. Subjects must have an ECOG performance status of 2 or less (see Appendix1).
4. Subjects must have a life expectancy of at least 4 weeks.
5. Subjects must be able to consume oral medication.
6. Subjects must have recovered from the toxic effects of any prior chemotherapy to =< Grade 1 (except alopecia).
7. Required initial laboratory values:

   1. Creatinine ≤ 2.0mg/dL
   2. total or direct bilirubin ≤ 1.5mg/dL; SGPT (ALT) ≤ 3xULN
   3. negative pregnancy test for women with child-bearing potential.
8. Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
9. Subjects must have a left ventricular ejection fraction (LVEF) of ≥ 45%.

Exclusion Criteria:

1. Subjects with FAB M3 (t (15; 17) (q22; q21) [PML-RARα]) are not eligible.
2. Subjects must not be receiving any chemotherapy agents (except Hydroxyurea).

   a) Intrathecal methotrexate and cytarabine are permissible.
3. Subjects must not be receiving growth factors, except for erythropoietin.
4. Subjects with a "currently active" second malignancy, other than non-melanoma skin cancers are not eligible.
5. Subjects with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, myocardial infarction within the past 6 months or serious uncontrolled cardiac arrhythmia are not eligible.
6. Subjects taking the following are not eligible:

   1. Carbamazepine (e.g., Tegretol)
   2. Rifabutin (e.g., Mycobutin) or
   3. Rifampin (e.g., Rifadin)
   4. Rifapentine (e.g., Priftin)
   5. St. John's wort
   6. Clarithromycin (e.g., Biaxin)
   7. Cyclosporine (e.g. Neoral or Sandimmune)
   8. Diltiazem (e.g., Cardizem)
   9. Erythromycin (e.g., Akne-Mycin, Ery-Tab)
   10. Itraconazole (e.g., Sporanox)
   11. Ketoconazole (e.g., Nizoral)
   12. Telithromycin (e.g., Ketek)
   13. Verapamil (e.g., Calan SR, Isoptin, Verelan)
   14. Voriconazole (e.g., VFEND)
   15. Tacrolimus (e.g. Prograf) Subjects taking fluconozole, voriconizole, itraconazole, posaconazole, and ketokonazole within 72 hours of study drug starting are not eligible. Reinstitution of fluconozole, voriconizole, itraconazole, posaconazole, ketokonazole and diltiazem is permissible 72 hours after the last dose of sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Biochemical response | Baseline to day 4
  Defined by change in phosphorylated ribosomal protein S6 (pS6) positive blasts, measured as the % reduction in pS6 positive blasts from baseline to day 4. Biochemical response will be described by mean, median, standard deviation, range and coefficient of variation. The association between biochemical response and clinical response will be tested by Fisher's exact test.
Clinical response | Day 45
  Based on hematologic recovery/day 45 marrow assessed according to International Working Group (IWG) criteria. The association between biochemical response and clinical response will be tested by Fisher's exact test.
Incidence of adverse events | Up to day 45
  Recorded and graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Worse toxicity grades observed during treatment will be described. Toxicities will be graded and tabled.

SECONDARY OUTCOMES:
Overall response rate (ORR) (complete response [CR], CR with incomplete platelet recovery [CRp], or partial response) | Day 45
  Fraction of patients who achieve CR, CRp, or PR will be assessed. ORR and 95% exact confidence interval will be computed for all patients and for sensitive and resistant subgroups.
Relapse free survival (RFS) | Time from study entry to first documented progression, death, or last contact, assessed up to 2 years
  RFS will be estimated by the Kaplan-Meier method. A landmark analysis of RFS by clinical response (CR+CRp, CRi, PR or no response [NR]) will be computed from day 45 marrow assessment. Median values and 95% confidence intervals will be calculated.
Overall survival (OS) | Time from study entry to death or last contact, assessed up to 2 years
  OS will be estimated by the Kaplan-Meier method. A landmark analysis of RFS by clinical response (CR+CRp, CRi, PR or NR) will be computed from day 45 marrow assessment. Median values and 95% confidence intervals will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/